CLINICAL TRIAL: NCT02592096
Title: A Single Dose Phase I Clinical Study of Pazufloxacin Mesilate Ear Drops for the Patients With Otitis Media
Brief Title: Pazufloxacin Mesilate Ear Drops Clinical Trial Protocol
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zhaoke-2015-01
Record Dates: First submitted 2015-07-15; First posted 2015-10-30 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Otitis Media
Keywords: safety and bioavailability
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0.1% Pazufloxacin Mesilate Ear Drops (Experimental): 10 drips for ear dropping, 10 minutes for ear bath
  Interventions: Drug: 0.1% Pazufloxacin Mesilate Ear Drops
- 0.3% Pazufloxacin Mesilate Ear Drops (Experimental): 10 drips for ear dropping, 10 minutes for ear bath
  Interventions: Drug: 0.3% Pazufloxacin Mesilate Ear Drops
- 0.5% Pazufloxacin Mesilate Ear Drops (Experimental): 10 drips for ear dropping, 10 minutes for ear bath
  Interventions: Drug: 0.5% Pazufloxacin Mesilate Ear Drops
- Pazufloxacin mesilate injection (Active Comparator): 0.3g, 30 minutes for ventricular injection
  Interventions: Drug: Pazufloxacin mesilate injection

INTERVENTIONS:
Drug: 0.1% Pazufloxacin Mesilate Ear Drops
  Arms: 0.1% Pazufloxacin Mesilate Ear Drops
Drug: 0.3% Pazufloxacin Mesilate Ear Drops
  Arms: 0.3% Pazufloxacin Mesilate Ear Drops
Drug: 0.5% Pazufloxacin Mesilate Ear Drops
  Arms: 0.5% Pazufloxacin Mesilate Ear Drops
Drug: Pazufloxacin mesilate injection
  Arms: Pazufloxacin mesilate injection

SUMMARY:
To investigate the safety, tolerance, dynamic percolation model of single dose usage pazufloxacin mesilate ear drops for patients with acute suppurative otitis media or chronic suppurative otitis media

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years old, both gender;
2. Patients with acute or chronic suppurative otitis media, need to be treated partially by antimicrobial agents;
3. Written informed consent form.

Exclusion Criteria:

1. Allergic to quinolones antibiotics or severe allergic constitution;
2. Not able to collect otorrhea during the trial;
3. High severity with the need of combined antibiotics treatment;
4. Induced by pathogens, e.g.: fungus, virus (myringitis bullosa);
5. Combined otitis externa (e.g.: ear cellulitis, mumps), intracranial or extracranial complication (meningitis, cerebral abscess, thrombophlebitis of sigmoid sinus, Bezold's abscess, ear subperiosteal abscess);
6. Severe disease of cerebral, cardiopulmonary, renal hepatic, circulatory system;
7. Life-threatening disease, e.g.: malignant tumor or AIDS.
8. Renal hepatic dysfunction (ALT, AST ≥ 1.5 times of normal maximum level, Cr > normal maximum level);
9. Confirmed or suspected of alcohol/drug abuse record;
10. Neurological or psychiatric disease leading to inability of cooperation or not willing to follow the protocol or instruction;
11. Feminine patients who are in gestational, lactation period or having a birth plan in short-term;
12. Enrolled into other clinical trial in the past 3 months;
13. Not suitable for this trial according to investigator's judgment;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
safety and tolerance of pazufloxacin mesilate ear drops | 24 hours
  Any changes in vital signs; AE/SAE number

SECONDARY OUTCOMES:
PK of pazufloxacin mesilate ear drops | 24 hours
  blood samples will be collected at 0, 0.5, and one of the followed time points 2, 4, 6, 8 hours. AUC will be calculated based on the pazufloxacin mesilate concentration at above timepoints in blood.
PK of pazufloxacin mesilate ear drops | 24 hours
  blood samples will be collected at 0, 0.5, and one of the followed time points 2, 4, 6, 8 hours. Cmax will be calculated based on the pazufloxacin mesilate concentration at above timepoints in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Cue, MD, Principal Investigator — Qingdao Municipal Hospital
Locations (1):
- Qingdao Municipal Hospital, Qingdao, China